CLINICAL TRIAL: NCT04989010
Title: Safety Study of 89Zr-Anti-CLDN18.2 mAbs PET-CT Imaging in Patients With CLDN18.2 Positive Solid Tumors
Brief Title: Safety Study of 89Zr-Anti-CLDN18.2 mAbs PET Imaging in Patients With CLDN18.2 Positive Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS-CLDN18.2 001
Record Dates: First submitted 2021-07-20; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-NY005 injection (Experimental): Patients will receive a tracer (10 mg, IV) dose of Zr-89 (2-3 mCi) labeled anti-CLDN18.2 mAbs (89Zr-NY005)
  Interventions: Drug: 89Zr-NY005

INTERVENTIONS:
Drug: 89Zr-NY005 — 89Zr-NY005 injection followed by 89Zr-NY005 PET scan

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 89Zr-labeled anti-CLDN18.2 mAbs (89Zr-NY005) PET imaging in patients with CLDN18.2 positive solid tumors.

DETAILED DESCRIPTION:
After being fully informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Patients will receive an injection of anti-CLDN18.2 mAbs(89Zr-NY005) and will undergo PET/CT scanning to determine uptake of 89Zr-NY005 in tumor lesions and normal tissues and organs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent, and be able to complete the trial according to the requirement of the scheme;
2. Aged 18-80, male or female;
3. The clinical diagnosis was gastric cancer, esophageal cancer and pancreatic cancer;
4. Patients with biopsy-proven CLDN18.2 positive;
5. Patients diagnosed with solid tumors confirmed by histopathology or cytology test;
6. At least two measurable solid lesions has been examined by 18F-FDG PET/CT (RECIST1.1 standard);
7. ECOG score ≤ 0~3; Life expectancy of at least 3 months;
8. ALT, AST shall not exceed 3 times of the normal upper limit; Bun, Cr not exceed 1.5 times of the normal upper limit.
9. Other routine examinations are within the normal range or considered acceptable by the researchers.

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with systemic or locally severe infections, or other serious coexisting diseases;
3. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
4. Patients with autoimmune diseases, including rheumatoid arthritis;
5. Inadequate control of arrhythmias, including atrial fibrillation;
6. Uncontrolled hypertension;
7. Patients with allergies or allergies to any component of the imaging agent or antibody;
8. Patients who cannot undergo PET/CT imaging scan;
9. Syphilis, HBV, HCV, or HIV positive subjects;
10. Male and female subjects of reproductive age cannot take effective contraceptive measures;
11. Pregnant or lactating women;
12. Patients with a history of mental illness or related conditions;
13. Other subjects considered unsuitable by researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 89Zr-Anti-CLDN18.2 mAbs(NY005) | 1 year
  Biodistribution of 89Zr-Anti-CLDN18.2 mAbs (NY005) evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 89Zr-PET scans will be reported.
Pharmacokinetic analysis of 89Zr-Anti-CLDN18.2 mAbs (NY005). | 1 year
  Area under the radioactivity (SUVs) versus time (time from injection) curve (AUC) will be derived by integration and reported.
  Other pharmacokinetic parameters including peak radioactive uptake (Cmax) and time (Tmax) in different organs, clearance and volume of distribution, evaluated using a biexponential model and non-compartmental analysis, will be reported.
Dosimetry estimates of 89Zr-Anti-CLDN18.2 mAbs (NY005). | 1 year
  Absorbed dose (radioactive uptake) estimates for different organs and tissues calculated with the AUCs and the OLINDA/EXM dosimetry program will be obtained and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi No. 4 People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No